CLINICAL TRIAL: NCT03457441
Title: Evaluation of Near Visual Acuity With ODYSIGHT, a Smartphone Based Medical Application in Comparison to a Standardized Method
Brief Title: Evaluation of Near Visual Acuity With ODYSIGHT, a Smartphone Based Medical App in Comparison to a Standardized Method
Acronym: TIL-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tilak Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-A03250-53
Record Dates: First submitted 2018-02-20; First posted 2018-03-07 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Near Vision
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Near visual acuity +1.0 and +0.7 logMAR (Other): Subjects with near visual acuity between +1.0 and +0.7 logMAR , when eligible and providing informed consent, assigned to evaluation with OdySight mobile medical application
  Interventions: Other: Standards vision tests; Device: OdySight medical application assessment
- Near visual acuity +0.6 and +0.3 logMAR (Other): Subjects with near visual acuity between +0.6 and +0.3 logMAR , when eligible and providing informed consent, assigned to evaluation with OdySight mobile medical application
  Interventions: Other: Standards vision tests; Device: OdySight medical application assessment
- Near visual acuity +0.2 and +0.0 logMAR (Other): Subjects with near visual acuity between +0.2 and +0.0 logMAR , when eligible and providing informed consent, assigned to evaluation with OdySight mobile medical application
  Interventions: Other: Standards vision tests; Device: OdySight medical application assessment

INTERVENTIONS:
Other: Standards vision tests — Subjects vision : near visual acuity, contrast sensitivity and scotoma and metamorphopsia detection will be assessed by gold-standard tests and with the OdySight medical application
Device: OdySight medical application assessment — Subjects vision : near visual acuity, contrast sensitivity and scotoma and metamorphopsia detection will be assessed by gold-standard tests and with the OdySight medical application

SUMMARY:
This study evaluates the level of agreement between visual parameters tested using OdySight, a mobile application, and standards in office methods.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to correctly distinguish the body laterality (left and right)
* Able to recognize alphabet letters and read French
* Affiliated to or beneficiary of the French health care system
* Signed/written informed consent
* Subject presenting a level of visual acuity of one of his eyes that fits to one of the pre-set cohort (visual acuity between +1.0 and +0.7 logMAR, between +0.6 and +0.3 logMAR or between +0.2 and 0.0 logMAR); the two eyes can be included in two different cohorts.

Exclusion Criteria:

* Any pathology that is considered by the investigator as capable of affecting the quality of the main evaluation criteria.
* Pregnant and breastfeeding women.
* Subject not considered by the investigator or designee to correctly use OdySight modules after the training session

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
Near visual acuity assessment with OdySight versus with near visual acuity chart | 1 day ( During evaluation visit)
  To assess the equivalence between a smartphone based evaluation of near visual acuity with ODYSIGHT (NVA module) and a standardized method (Sloan ETDRS near vision letter chart).

SECONDARY OUTCOMES:
Near visual acuity assessment with OdySight versus with ETDRS chart | 1 day ( During evaluation visit)
  To assess the relation between the ETDRS visual acuity at a 4-meter distance and near visual acuity evaluated with ODYSIGHT (NVA module)

OTHER OUTCOMES:
Contrast sensitivity assessment with OdySight versus with Pelli-Robson | 1 day ( During evaluation visit)
  To compare the smartphone based evaluation of the contrast sensitivity with ODYSIGHT (contrast sensitivity module) and a standardized method (Pelli-Robson chart)
Scotoma/metamorphopsia detection with OdySight versus with standard Amsler grid | 1 day ( During evaluation visit)
  To compare the smartphone based evaluation of the Amsler Grid with ODYSIGHT (Amsler grid module) and standardized methods (paper Amsler Grid)
Global functional disorders assessment with Odysight versus with OCT | 1 day ( During evaluation visit)
  To compare functional disorder(s) detected or measured by ODYSIGHT application with anatomical data (OCT: Optical coherence tomography)

CONTACTS AND LOCATIONS:
Overall Officials: Saddek Mohan-Saïd, MD, Principal Investigator — Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts
Locations (1):
- Centre Hospitalier National d'Ophtahlomogie du Quinze-Vingts, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brucker J, Bhatia V, Sahel JA, Girmens JF, Mohand-Said S. Odysight: A Mobile Medical Application Designed for Remote Monitoring-A Prospective Study Comparison with Standard Clinical Eye Tests. Ophthalmol Ther. 2019 Sep;8(3):461-476. doi: 10.1007/s40123-019-0203-9. Epub 2019 Jul 25. PMID 31346977